CLINICAL TRIAL: NCT07402759
Title: Impact of tdrd9 Gene Mutations in the Therapeutic Response to L-carnitine in Oligoasthenozoospermic Men
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: South Valley University (Other)
Responsible Party: Principal Investigator, Mostafa Abd-Elhakeem Ameen, Resident at dermatology, venereology and andrology department south valley university hospital, principal investigator, South Valley University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Svu-med-dva021-4-25-12-5
Record Dates: First submitted 2026-01-18; First posted 2026-02-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Oligoasthenozoospermia; Male Infertility
Keywords: Tdrd9; L-carnitine; Sperm motility; Semen analysis; Total motile sperm count
MeSH Terms: conditions — Infertility, Male | interventions — Carnitine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Tdrd9 positive and negative (Experimental): L-carnitine
  Interventions: Drug: L-carnitine

INTERVENTIONS:
Drug: L-carnitine — Dietary supplement

SUMMARY:
Infertility remains a significant global burden. Estimates suggest that 10-15% of couples worldwide experience infertility, with male infertility being the underlying cause in 20-50% of cases. For the majority of cases however the etiology remains unknown, and is termed idiopathic infertility. Azoospermia, absence of spermatozoa in the semen, is one of the most common reasons for infertility in men, with a prevalence of 1% in the general population, and over 15% in infertile men.

Oligozoospermia is a major cause of male infertility, yet its genetic basis remains partially understood. Oligozoospermia refers to sperm concentrations below established reference limits (e.g. 16 million/ml, 95% confidence interval 15-18 million/ml; WHO 2021).

Numerous studies have demonstrated a strong genetic basis for oligozoospermia, with genetic abnormalities, such as abnormalities in chromosome number or structure, azoospermia factor region (AZF) deletion on the Y chromosome and cystic fbrosis transmembrane conduction regulator (CFTR) gene mutations, reported in men with otherwise unexplained oligozoospermia and azoospermia. Moreover, previous studies have identifed more than 400 genes that are specifcally or potentially associated with fertility regulation while potentially contributing to the widespread genetic heterogeneity associated with dyszoospermia. For example, mutations in RPL10L and MAGEB have been reported to cause oligozoospermia. However, mutations in only a few genes have been shown to cause male infertility, and the candidate pathogenic genes for oligozoospermia still need to be studied further.

Recent studies have implicated the Tudor Domain Containing 9 (TDRD9) gene in the regulation of spermatogenesis through its role in piRNA pathway and transposon silencing. A 2024 study identified compound heterozygous mutations-c.1115+3A>G (splicing variant) and c.958delC (frameshift variant)-in a Chinese family with idiopathic oligozoospermia, resulting in aberrant splicing and truncated TDRD9 protein products.

Tudor domain-containing protein 9 (TDRD9) is an RNA helicase that is highly expressed in germlines. TDRD9 expression has been detected in mitotic spermatogonia, meiotic spermatocytes and haploid spermatids in the testis. In male infertility cases, TDRD9 has been reported to be involved in the silencing of long intersperm-1 retrotransposons, suggesting an association between TDRD9 mutations and non-obstructive azoospermia.

TDRD9 is implicated in spermatogenesis and piRNA pathway integrity. Variants may affect sperm quality and response to treatments. L-carnitine is widely used as an antioxidant and metabolic supplement shown to improve sperm parameters in some infertile men. This study will test whether TDRD9 mutation status predicts therapeutic benefit from L-carnitine.

DETAILED DESCRIPTION:
Genetic Basis of Male Infertility with Emphasis on Oligozoospermia and the Role of TDRD9 Infertility represents a major global health concern, affecting approximately 10-15% of couples worldwide. Male factors contribute to infertility in nearly 20-50% of these cases, either as an isolated cause or in combination with female factors. Despite advances in diagnostic techniques, the etiology of male infertility remains unidentified in a substantial proportion of patients and is therefore classified as idiopathic infertility. Among the various causes of male infertility, abnormalities in sperm production and function constitute the most frequent underlying pathology.

Azoospermia, defined as the complete absence of spermatozoa in the ejaculate, is one of the most severe manifestations of male infertility. It affects approximately 1% of the general male population and accounts for more than 15% of infertility cases among men. Azoospermia may be obstructive or non-obstructive, with the latter reflecting intrinsic defects in spermatogenesis and frequently having a genetic basis.

Oligozoospermia, characterized by reduced sperm concentration, is another major contributor to male infertility and often represents a milder but clinically significant spermatogenic failure. According to the World Health Organization (WHO) 2021 reference values, oligozoospermia is defined as a sperm concentration below 16 million spermatozoa per milliliter (95% confidence interval: 15-18 million/mL). Although environmental, lifestyle, endocrine, and infectious factors have been implicated, accumulating evidence indicates that oligozoospermia has a strong genetic component. Nevertheless, its molecular and genetic underpinnings remain only partially understood.

Genetic Abnormalities in Oligozoospermia and Azoospermia Genetic defects are increasingly recognized as major contributors to otherwise unexplained oligozoospermia and azoospermia. Classical genetic abnormalities include numerical and structural chromosomal anomalies, such as Klinefelter syndrome (47,XXY), balanced translocations, and inversions. Microdeletions within the azoospermia factor (AZF) regions of the Y chromosome (AZFa, AZFb, and AZFc) are among the most well-established genetic causes of impaired spermatogenesis. In addition, mutations in the cystic fibrosis transmembrane conductance regulator (CFTR) gene are commonly associated with congenital bilateral absence of the vas deferens and obstructive azoospermia.

Beyond these well-characterized abnormalities, next-generation sequencing technologies have enabled the identification of hundreds of genes potentially involved in spermatogenesis. To date, more than 400 genes have been reported to be specifically or potentially associated with male fertility regulation, reflecting the remarkable genetic heterogeneity underlying dyszoospermia. Mutations in genes such as RPL10L, which plays a role in ribosomal function during spermatogenesis, and MAGEB, involved in germ cell development, have been implicated in oligozoospermia. However, despite these discoveries, pathogenic variants in only a limited number of genes have been conclusively linked to male infertility, highlighting the need for continued investigation into novel candidate genes.

TDRD9 and Its Role in Spermatogenesis Recent studies have highlighted the Tudor Domain Containing 9 (TDRD9) gene as a critical regulator of spermatogenesis. TDRD9 encodes a germline-specific RNA helicase that plays an essential role in the PIWI-interacting RNA (piRNA) pathway, a key defense mechanism that suppresses transposable elements during germ cell development. Proper transposon silencing is crucial for maintaining genomic stability in germ cells, and disruption of this process can lead to impaired spermatogenesis and infertility.

TDRD9 is highly expressed in the testis, with expression detected across multiple stages of germ cell development, including mitotic spermatogonia, meiotic spermatocytes, and haploid spermatids. Functional studies have demonstrated that TDRD9 participates in the silencing of long interspersed nuclear element-1 (LINE-1) retrotransposons, thereby protecting germ cell integrity. Defects in this pathway have been associated with spermatogenic arrest and non-obstructive azoospermia.

A recent 2024 study provided compelling clinical evidence for the involvement of TDRD9 in human male infertility. In a Chinese family with idiopathic oligozoospermia, compound heterozygous mutations in TDRD9-namely a splice-site variant (c.1115+3A>G) and a frameshift variant (c.958delC)-were identified. These mutations resulted in aberrant mRNA splicing and truncated protein products, leading to impaired TDRD9 function. This study strengthened the causal link between TDRD9 dysfunction and defective spermatogenesis and expanded the spectrum of genes implicated in oligozoospermia.

ELIGIBILITY:
Inclusion Criteria Male participants aged 20-50 years

Clinical diagnosis of oligoasthenozoospermia, confirmed by two semen analyses according to WHO 2010/2021 criteria:

Sperm concentration <15 million/mL, and Progressive motility <32% Attempting conception with a partner for ≥12 months, or referred for infertility evaluation Willing and able to take oral L-carnitine and comply with all study visits and procedures Able and willing to provide written informed consent, including consent for genetic testing (TDRD9 analysis) Exclusion Criteria Known obstructive azoospermia Grade III varicocele requiring surgical correction, unless repaired ≥6 months prior to enrollment Use of fertility supplements or hormonal therapy within the 3 months prior to enrollment (washout required) Active genitourinary infection (e.g., prostatitis) or systemic illness known to affect fertility Known severe systemic disease, including uncontrolled diabetes mellitus or severe hepatic or renal disease Known hypersensitivity or allergy to L-carnitine History of testicular cancer or receipt of chemotherapy within the past 2 years

Ages: 20 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2026-01-01 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Change in total motile sperm count (TMSC) from baseline to 3 months | Baseline to 3 months
  Total motile sperm count (TMSC), calculated as semen volume × sperm concentration × percentage of progressively motile sperm, measured at baseline and after 3 months of oral L-carnitine therapy. The outcome is expressed as the mean change in TMSC (million motile sperm per ejaculate) from baseline to 3 months and compared between men with and without TDRD9 gene mutations.
  Unit of Measure:
  Million motile sperm per ejaculate

SECONDARY OUTCOMES:
Change in sperm concentration from baseline to 3 months | Baseline to 3 months
  Sperm concentration measured by semen analysis according to WHO criteria at baseline and after 3 months of treatment. Outcome is the mean change in sperm concentration (million/mL) from baseline to 3 months, compared between TDRD9 mutation carriers and non-carriers.
  Unit of Measure:
  Million sperm per mL
Change in normal sperm morphology from baseline to 3 months | Baseline to 3 months
  Percentage of sperm with normal morphology assessed using strict WHO criteria at baseline and after 3 months. Outcome is the mean change in normal morphology (%) from baseline to 3 months between groups.
  Unit of Measure:
  Percentage (%)
Change in semen volume from baseline to 3 months | Baseline to 3 months
  Semen volume measured in milliliters at baseline and after 3 months of treatment. Outcome is the mean change in semen volume (mL) from baseline to 3 months.
  Unit of Measure:
  Milliliters (mL)
Change in serum follicle-stimulating hormone (FSH) levels from baseline to 3 months | Baseline to 3 months
  Serum FSH measured at baseline and after 3 months of therapy. Outcome is the mean change in FSH level (IU/L) from baseline to 3 months.
  Unit of Measure:
  IU/L

CONTACTS AND LOCATIONS:
Overall Officials: Eisa Mohammed Hegazy, Study Director — South Valley University; Mahmoud Ahmed Ali, Assistant professor, Study Chair — Aswan University Hospital
Locations (1):
- Qena university hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lahimer M, Gherissi O, Ben Salem N, Ben Mustapha H, Bach V, Khorsi-Cauet H, Khairi H, Ben Ali H, BenKhalifa M, Ajina M. Effect of micronutrients and L-carnitine as antioxidant on sperm parameters, genome integrity, and ICSI outcomes: randomized, double-blind, and placebo-controlled clinical trial. Antioxidants. 2023 Oct 31;12(11):1937.
- [Background] Okutman O, et al. A no-stop mutation in MAGEB4 is a possible cause of rare X-linked azoospermia and oligozoospermia in a consanguineous Turkish family. J Assist Reprod Genet. 2017;34(5):683-94.
- [Background] Esteves SC. Who cares about oligozoospermia when we have ICSI. Reproductive biomedicine online. 2022 May 1;44(5):769-75.
- [Background] Wang W, Feng Y, Dong J, Zhou Z, Jing J, Li Z, Chen L, Lin X, Ma J, Yao B. A Novel Compound Heterozygous Mutation in TDRD9 Causes Oligozoospermia. Reproductive Sciences. 2024 Nov;31(11):3413-9.
- [Background] Babakhanzadeh E, Khodadadian A, Rostami S, Alipourfard I, Aghaei M, Nazari M, Hosseinnia M, Mehrjardi MY, Jamshidi Y, Ghasemi N. Testicular expression of TDRD1, TDRD5, TDRD9 and TDRD12 in azoospermia. BMC medical genetics. 2020 Dec; 21:1-7. rmia when we have ICSI. Reproductive biomedicine online. 2022 May 1;44(5):769-75.